CLINICAL TRIAL: NCT02428699
Title: Comparison of Plasma Levels of n-3 Fatty Acids After Ingestion of an Emulsified Cod Liver Oil Product and a Non Emulsified Cod Liver Oil Product
Brief Title: Study Comparing Blood Levels of Fatty Acids After Consuming Two Forms of Cod Liver Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202359
Record Dates: First submitted 2015-04-09; First posted 2015-04-29 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-06

CONDITIONS: Growth and Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): 30mL Test contains 10%w/w cod oil + 10%w/w cod liver oil in an emulsion formulation
  Interventions: Other: Emulsified cod liver oil product
- Control (Active Comparator): 5.8mL of cod liver oil in a free flowing non-emulsified formulation
  Interventions: Other: Non-emulsified cod liver oil product

INTERVENTIONS:
Other: Emulsified cod liver oil product — Participants are required to consume the dose (30 mL) within 1 min, followed by up to 300 mL of apple juice which needs to be consumed within 2 min
  Arms: Test
Other: Non-emulsified cod liver oil product — Participants are required to consume the dose (5.8 mL) within 1 min, followed by up to 300 mL of apple juice which needs to be consumed within 2 min
  Arms: Control

SUMMARY:
This study is designed to compare the incremental area under the curve from 0 to 24h (iAUC0-24h) of plasma levels of n-3 fatty acids (sum of total and free eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) after ingestion of an emulsified product and a non-emulsified reference control of free flowing cod liver oil at the lowest appropriate dose that is practically acceptable, and as near as possible to the test products' recommended daily dose.

DETAILED DESCRIPTION:
Many dietary lipids are in the form of triglycerides, ethyl esters or phospholipids. During digestion these lipids are subject to hydrolysis, in particular by pancreatic triglyceride lipase. To facilitate the action of the enzyme, lipids are emulsified by the action of bile salts. By increasing the surface area of the fat globules, emulsification increases access to the lipids by pancreatic triglyceride lipase. This study is designed to compare iAUC0-24h of plasma levels of n-3 fatty acids (sum of total and free EPA and DHA) after ingestion of an emulsified product and a non-emulsified reference control of free flowing cod liver oil at the lowest appropriate dose that is practically acceptable, and as near as possible to the test products' recommended daily dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 45 years (both inclusive)
* Body mass index (BMI) of 18.5-29.9 kg/m2 inclusive

Exclusion Criteria:

* Pregnant or lactating women
* Allergy/intolerance to any study material
* Current or recurrent disease, within 12 months of screening that could affect the metabolism of drug
* Participants who have taken any drug known to induce or inhibit hepatic drug metabolism in 30 days prior to screening
* Positive serum Hepatitis B surface antigen, Hepatitis C antibodies or Human Immunodeficiency Virus (HIV), alcohol or drug abuse
* Smokers taking >5 cigarettes/day; prior or current use of any other nicotine containing product
* Blood donated within 3 months of screening
* Consumed n-3 rich food or beverage or n-3 fortified food or beverage within 72h prior to each study session

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Conus N, Burgher-Kennedy N, van den Berg F, Kaur Datta G. A randomized trial comparing omega-3 fatty acid plasma levels after ingestion of emulsified and non-emulsified cod liver oil formulations. Curr Med Res Opin. 2019 Apr;35(4):587-593. doi: 10.1080/03007995.2018.1512479. Epub 2018 Sep 28. PMID 30106311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one Centre in United Kingdom.
Pre-assignment Details: A total of 93 participants were screened, out of which 50 participants were randomized. 39 participants failed screening and 2 participants withdrew from the study. 2 participants discontinued due to other reasons (reason not specified).
Groups:
- Scott's Emulsion Followed by Non Emulsified Cod Liver Oil: Sequence 1: Participants were administered 30 milliliters (mL) of Scott's emulsion (10 percent [%] Cod Liver Oil, 10% Cod Oil) followed by 300 mL of apple juice in period 1. After a washout period of 2 weeks participants were administered 5.8 mL non emulsified cod liver oil, followed by 300 ml apple juice in period 2.
- Non Emulsified Cod Liver Oil Followed by Scott's Emulsion: Sequence 2: Firstly, participants were administered 5.8 mL non emulsified cod liver oil, followed by 300 mL of apple juice in Period 1. After a washout period of 2 weeks participants were administered test product i.e. 30 mL of Scott's emulsion (10 % Cod Liver Oil, 10% Cod Oil) followed by 300 mL apple juice in period 2.
Period: Period 1
Arm/Group | Scott's Emulsion Followed by Non Emulsified Cod Liver Oil | Non Emulsified Cod Liver Oil Followed by Scott's Emulsion
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Washout Period 1
Arm/Group | Scott's Emulsion Followed by Non Emulsified Cod Liver Oil | Non Emulsified Cod Liver Oil Followed by Scott's Emulsion
Started | 25 | 25
Completed | 24 | 23
Not Completed | 1 | 2
Not completed — Screen Failure | 1 | 2
Period: Period 2
Arm/Group | Scott's Emulsion Followed by Non Emulsified Cod Liver Oil | Non Emulsified Cod Liver Oil Followed by Scott's Emulsion
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (N=50) was analysis population, defined as all participants who were randomized and administered at least one study treatment during the study.
Groups:
- Overall Study: Test product : 30 mL Scott's Emulsion containing 10% Cod Liver Oil, 10% Cod Oil. Reference product: 5.8 mL of non emulsified free flowing cod liver oil
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incremental Area Under the Curve to 24 Hours (h) (iAUC0-24h) of the Sum of Plasma Total and Free n-3 Fatty Acids (Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA)
Description: The AUC was calculated using the trapezoidal method and using nominal time points from 0, 2, 4, 6, 8, 10, 12 and 24 h respectively. The AUC was divided by the total duration to represent a weighted mean incremental change over time. Higher values of AUC demonstrate better rate of absorption over time than lower values.
Time Frame: Baseline and up to Day 2
Population: Per protocol (PP) population (N=47) was the primary population of analysis defined as all participants in the safety population who have at least one post-baseline assessment of efficacy considered unaffected by protocol violations. From the PP population, 3 participants were not analysed in test group and 2 in control group, due to missing data.
Measure: Mean (Standard Deviation); unit: Microgram per mililiter (µg/mL)
Groups:
- Test Product: 30 mL Scott's emulsion containing 10% cod liver Oil, and 10% cod oil
- Reference Product: 5.8 mL of non emulsified free flowing cod liver oil
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
Microgram per mililiter (µg/mL) | 13.19 (8.368) | 7.73 (6.532)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Superiority; p < .0001, ANCOVA; Subject as random effect,treatment and period as fixed effects,subject and period level baseline values for plasma total and free acids as covariates; Mean Difference (Net) = 5.16, 95% CI 2-sided [2.79 to 7.53] — Difference is test minus reference such that a positive difference favors the test treatment

2. Secondary Outcome: iAUC0-24h of Sum of Total and Free DHA
Description: as for outcome 1
Time Frame: Baseline and up to Day 2
Population: PP population (N=47) was the primary population of analysis defined as all participants in the safety population who have at least one post-baseline assessment of efficacy considered unaffected by protocol violations. From the PP population, 3 participants were not analysed in test group and 2 in control group, due to missing data.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 5.09 (6.118) | 2.89 (4.225)

3. Secondary Outcome: iAUC0-24h of Sum of Total and Free EPA
Description: as for outcome 1
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 8.10 (2.810) | 4.84 (2.903)

4. Secondary Outcome: iAUC0-10h of Sum of Total and Free DHA
Description: The AUC was calculated using the trapezoidal method and using nominal time points from 0, 2, 4, 6, 8, and 10h respectively. The AUC was divided by the total duration to represent a weighted mean incremental change over time. Higher values of AUC demonstrate better rate of absorption over time than lower values.
Time Frame: Upto 10 h
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 7.51 (6.810) | 3.86 (4.011)

5. Secondary Outcome: iAUC0-10h of Sum of Total and Free EPA
Description: as for outcome 4
Time Frame: Upto 10 h
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Test Product: 30 mL Scott's Emulsion containing 10% Cod Liver Oil, 10% Cod Oil
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 7.28 (2.893) | 3.97 (2.493)

6. Secondary Outcome: iAUC0-10h of Sum of Total and Free DHA and EPA
Description: as for outcome 4
Time Frame: Upto 10 h
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 14.79 (9.336) | 7.83 (6.133)

7. Secondary Outcome: Maximum Concentration (Cmax) of Sum of Total and Free DHA and EPA
Description: Blood sampleswere taken at time points 0,2,4,6,8,10,12 and 24h. Maximum plasma concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 98.37 (26.595) | 90.48 (26.252)

8. Secondary Outcome: Cmax of Sum of Total and Free DHA
Description: Blood samples were taken at time points 0,2,4,6,8,10,12 and 24h. Maximum plasma concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 70.61 (19.698) | 64.73 (19.229)

9. Secondary Outcome: Cmax of Sum of Total and Free EPA
Description: Blood sampleswere taken at time points 0,2,4,6,8,10,12 and 24h. Maximum plasma concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
µg/mL | 28.89 (8.205) | 26.27 (8.894)

10. Secondary Outcome: Time to Maximum Concentration (Tmax) of Sum of Total and Free DHA and EPA
Description: Blood samples will be taken at time points 0,2,4,6,8,10,12 and 24h. Time to maximum concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
h | 5.77 (2.208) | 7.73 (3.480)

11. Secondary Outcome: Tmax of Sum of Total and Free DHA
Description: Blood samples will be taken at time points 0,2,4,6,8,10,12 and 24h. Time to maximum concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
h | 5.23 (1.790) | 7.56 (4.219)

12. Secondary Outcome: Tmax of Sum of Total and Free EPA
Description: Blood samples will be taken at time points 0,2,4,6,8,10,12 and 24h.Time to maximum concentration was determined.
Time Frame: Baseline and up to Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 44 | 45
h | 8.36 (4.979) | 8.00 (3.464)

ADVERSE EVENTS:
Time Frame: approximately 45 days
Description: Safety population (N=50) included all participants who were randomized and administered at least one study treatment during the study (47 participants were treated with both Scott's Emulsion Original and Cod liver oil; 1 participant was treated with Scott's Emulsion only and 2 were treated with Cod liver oil only). Therefore, a total of 48 participants were included in Scotts emulsion (test product) arm and 49 in Cod liver oil (reference product) arm.
Arm/Group | Test Product | Reference Product
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 9/48 | 3/49
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=48) | Reference Product (N=49)
Headache (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.